CLINICAL TRIAL: NCT02425280
Title: How to Help War-affected Children and Adolescents: the Role of Memory Functions in Therapeutic Intervention
Brief Title: Effectiveness of Narrative Exposure Therapy Among Refugee Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Kirsi Peltonen, Postdoctoral Researcher, Tampere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 275804
Record Dates: First submitted 2015-04-15; First posted 2015-04-23 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Narrative Exposure Therapy; Treatment as Usual
MeSH Terms: interventions — Therapeutics

ARMS (2):
- Narrative Exposure Therapy (Experimental): For the intervention group receiving Narrative Exposure Therapy treatment, the intervention will last for approximately three months and include 10-12 weekly sessions of 60-90 minutes. The course of the intervention will follow the NET manual (Schauer et al., 2011).
  Interventions: Behavioral: Narrative Exposure Therapy
- Treatment as Usual (Active Comparator): For the TAU control group, participants will receive the usual care for posttraumatic stress symptoms currently offered by each unit.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy
  Arms: Narrative Exposure Therapy
Behavioral: Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
This study aims to understand how war trauma affects children's and adolescents' memory functions and mental health, and whether Narrative Exposure Therapy is effective in enhancing optimal memory functions and alleviating mental health problems. The study analyzes the mental health and cognitive and emotional healing mechanisms of therapeutic intervention among war-affected children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* 9-17 years old
* has spent some part of her/his life living in a country where organized violence was taking place, or at a refugee camp
* suffers from significant stress symptoms thought be trauma-related

Exclusion Criteria:

* acute psychosis
* intellectual disability

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Post-traumatic Stress as measured by Revised Impact of Event Scale | 9 months
Depression as measured by Depression Self-Rating Scale for Children | 9 months
Psychological Distress as measured by Strengths and Difficulties Questionnaire | 9 months
Resilience as measured by Child and Youth Resilience Measure | 9 months
Cognitive Performance as measured by Working Memory Test Battery for Children | 9 months

SECONDARY OUTCOMES:
Quality of Traumatic Memory as measured by Trauma Memory Quality Questionnaire | 9 months
Trauma Related Cognitions as measured by Children's Post Traumatic Cognitions Inventory | 9 months
General functioning of autobiographical memory as measured by reported life events | 9 months

OTHER OUTCOMES:
Subjective distress during therapy measured by Subjective Units of Distress Scale | 9 months
Peritraumatic Dissociation measured by Peritraumatic Dissociative Experiences Questionnaire | once, at baseline

CONTACTS AND LOCATIONS:
Locations (3):
- Finland (3):
  - Centre for Torture Survivors, Helsinki
  - Family Counselling Centre of the City of Tampere, Tampere
  - Psychiatric Clinic for Traumatized Children at Tampere University Hospital, Tampere

REFERENCES:
- [Derived] Kangaslampi S, Garoff F, Peltonen K. Narrative exposure therapy for immigrant children traumatized by war: study protocol for a randomized controlled trial of effectiveness and mechanisms of change. BMC Psychiatry. 2015 Jun 17;15:127. doi: 10.1186/s12888-015-0520-z. PMID 26081580